CLINICAL TRIAL: NCT01341548
Title: A Phase III, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group, Multicenter Evaluation of Civamide Nasal Solution 0.01% in the Prevention of Cluster Headaches During an Episodic Cluster Headache Period
Brief Title: Civamide Nasal Solution for Cluster Headache
Acronym: ECH
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WL-1001-02-06
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Episodic Cluster Headache
Keywords: Nasal; Cluster Headache; Episodic Cluster; Headache; Phase 3; Civamide; TRPV-1 Receptor
MeSH Terms: conditions — Cluster Headache; Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Civamide Nasal Solution 0.01% (Active Comparator)
  Interventions: Drug: Civamide nasal solution 0.01%
- Vehicle Solution (Placebo Comparator)
  Interventions: Drug: Civamide nasal solution 0.01%

INTERVENTIONS:
Drug: Civamide nasal solution 0.01% — 20ug/dose, BID for 7 days 0.1 ml to each nostril

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intranasally administered civamide nasal solution in the prevention of cluster headaches during an episodic cluster headache period.

DETAILED DESCRIPTION:
This is a double-blind, randomized, vehicle-controlled, parallel-group, multi-center, phase III efficacy and safety study of civamide nasal solution 0.01% in the prevention of cluster headaches during an episodic cluster headache period. Approximately 180 subjects (about 90 per treatment group),will be enrolled and randomized to double-blind treatment with either civamide nasal solution 0.01% or vehicle solution at approximately 50 study sites with about 2-5 subjects randomized per enrolling site.

This study consists of four periods beginning with a Screening Period, lasting for a minimum of 1 day to a maximum of 12 months, during which a subject previously diagnosed with episodic cluster headaches is not experiencing cluster headaches and is awaiting the onset of their next episodic cluster headache period and subsequent enrollment. The Screening Period is followed by a 31-day study, consisting of a 3-day Baseline Period which may begin with the onset of an episodic cluster headache period and ends on the day prior to initiating treatment (Day -1). Subjects return for Visit 2 (Day 1, Pre-Dose) and the Treatment Period begins, consisting of seven (7) days of double-blind treatment. The Treatment Period is immediately followed by a twenty-one (21) day Post-Treatment Observation Period.

ELIGIBILITY:
Inclusion Criteria:

* Written IRB-approved informed consent has been obtained and signed, within 12 months of entering into the Baseline Period (Day -3).
* Male or female 18 years or older.
* Subject has ≥2 year history of episodic cluster headache with at least 2 previous episodic cluster headache periods.
* Cluster Headaches must meet the following International Headache Society Diagnostic Criteria :

  * Severe, unilateral, orbital, superorbital and/or temporal pain lasting 15 to 180 minutes untreated.
  * Headache is associated with at least one of the following which have to be present on the side of the pain:

    * Conjunctival injection
    * Lacrimation
    * Nasal Congestion
    * Rhinorrhea
    * Forehead and facial sweating
    * Miosis
    * Ptosis
    * Eyelid edema or
    * A sense of restlessness or agitation
* The current episodic cluster headache period is expected to last at least 5 weeks but no more than 24 weeks from the time of entry into the Baseline Period (Day -3), based on the average duration of the subject's usual episodic cluster headache period.
* At least one cluster headache (but no more than 8) daily on each of the three days of the Baseline Period (Days -3, -2, -1) immediately preceding Study Day 1.
* The subject is in generally good health, other than history of episodic cluster headache.
* The subject agrees not to begin any new concurrent medications or restricted medications during their participation in study.
* All females of childbearing potential must have a negative urine and/or serum pregnancy test prior to entry into the Treatment Period.
* Females of childbearing potential agree to use an approved form of birth control or to abstain from sexual activity during the study.
* Subject can read and write in the local language and can be expected to reliably follow study procedures.

Exclusion Criteria:

* Clinical, historical or previous laboratory evidence of significant cardiovascular, renal, gastrointestinal, pulmonary, hepatic, endocrine, neurological (not including cluster headaches), psychological, or other systemic disease that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the subject.
* Presence of a significant nasal disorder.
* Initiation of a medication, discontinuation of a medication or a change in the regimen of existing medication(s) or therapies for prophylaxis of cluster headaches in the 17 days prior to entering the Treatment Period (Study Day 1).
* Use of systemic steroids to treat the current cluster headache episode.
* Use of restricted medications/treatments within the given time period prior to the Treatment Period and throughout the study (Table 1 of Protocol)
* Subject has difficulty distinguishing his/her episodic cluster headache attacks from other types of headaches, such as tension type headaches.
* Presence of chronic paroxysmal hemicrania, transformed migraine, or analgesic rebound headaches.
* Females who are pregnant, breast-feeding, or planning to become pregnant during the study.
* Subject has a history of alcohol and/or drug abuse within 12 months prior to the Screening Visit..
* Subject has known hypersensitivity to or contraindication to the use of civamide, capsaicin, or to any excipient of the clinical formulation.
* Subject has participated in another investigational study or taken another investigational drug within the past 4 weeks.
* Subject has participated in prior efficacy studies of intranasal civamide: WL-1001-02-01, WL-1001-02-02, WL-1001-02-03 or WL-1001-02-05. (This does not include any subject who entered the screening period for study WL-1001-02-01, WL-1001-02-02, WL-1001-02-03 or WL-1001-02-05 but did not randomize to treatment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The Percent Change in the Number of Cluster Headaches per Week from Baseline to Weeks 1 through 3 of the Post-Treatment Observation Period for the Modified Intent-to-Treat Population | Weeks 1 - 3 of the Post-Treatment Observation Period

SECONDARY OUTCOMES:
The Percent Change in the Number of Cluster Headaches per Week from Baseline to Weeks 1 through 3 of the Post-Treatment Observation Period for the Intent-to-Treat and Per Protocol Populations | Weeks 1 - 3 of the Post-Treatment Observation Period
The Percent Change in the Number of Cluster Headaches per Week from Baseline to Individual Weeks 1, 2, and 3 of the Post-Treatment Observation Period for the Modified Intent-to-Treat and the Per Protocol Populations | Individual Weeks 1, 2 and 3 of the Post-Treatment Observation Period
The Change in the Number of Cluster Headaches per Week from Baseline to Weeks 1 through 3 and to Individual Weeks 1, 2, and 3 for the Post-Treatment Observation Period for the Modified Intent-to-Treat and the Per Protocol Populations | Weeks 1 - 3 and to Individual Weeks 1, 2, and 3 for the Post-Treatment Observation Period

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, M.D., Study Director — Winston Laboratories

IPD SHARING:
Plan to Share IPD: No